CLINICAL TRIAL: NCT04204746
Title: The Effects of Different Fresh Gas Flows and Different Anesthetics on Airway Temperature and Moisture in Patients Who Underwent General Anesthesia
Brief Title: The Affecting Factors on Airway Temperature and Moisture
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ozkan Onal, Professor, Selcuk University
Other Study IDs: E.90598
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: General Anesthesia
Keywords: general anesthesia; fresh gas; moisture; temperature; respiratory circuit

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3 lt/min: Patients in the study were divided into two main groups according to the standard fresh gas flow administered (3-6 L/min). Each main group was then divided into subgroups as follows: sevoflurane + remifentanil, desflurane + remifentanil, or propofol + remifentanil (TIVA). These six groups were further divided into two groups according to use or non-use of a heat and moisture exchanger (HME) filter.
  Interventions: Other: We will observe and evaluate the temperature and moisture in the respiratory circuit by a thermo-hygrometer.
- 6 lt/min: Patients in the study were divided into two main groups according to the standard fresh gas flow administered (3-6 L/min). Each main group was then divided into subgroups as follows: sevoflurane + remifentanil, desflurane + remifentanil, or propofol + remifentanil (TIVA). These six groups were further divided into two groups according to use or non-use of a heat and moisture exchanger (HME) filter.
  Interventions: Other: We will observe and evaluate the temperature and moisture in the respiratory circuit by a thermo-hygrometer.

INTERVENTIONS:
Other: We will observe and evaluate the temperature and moisture in the respiratory circuit by a thermo-hygrometer.

SUMMARY:
There is no literature information about the flow rate of fresh gas mixture (air+O2) in the patients who underwent general anesthesia. Different flow rates of fresh gas mixture are used in both the investigator's hospital and the experiences of the anesthesiologists. It is aimed to study the effects of different fresh gas flow rates on the rate of temperature and moisture of the airway of patients who underwent general anesthesia.

DETAILED DESCRIPTION:
Under physiological conditions, inhaled air is heated and humidified as it passes through the nose and upper airways until reaching the alveoli. This mechanism is bypassed by endotracheal intubation. Ventilation with dry and cold compressed gases leads to loss of water and heat from the respiratory tract. Drying of the respiratory tract can lead to destruction of the cilia and mucous membranes, resulting in decreased mucociliary transport and increased concentration of secretions.There is no definitive literature on fresh gas mix (oxygen + air) flow rates in patients under general anesthesia. This study aimed to investigate whether two fresh gas flow rates routinely employed in the authors' practice affected airway temperature and humidity.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-65 years underwent general anesthesia -

Exclusion Criteria:admitted to emergency and trauma, history of advanced cardiac disease, cigarette use ≥ 3 packet/day, pulmonary parenchymal disease such as malignancy or chronic obstructive pulmonary disease (COPD), history of thyroid disease, body mass index (BMI) greater than 30 kg/m2, alcohol and substance addiction, mentally deficiency, pregnancy or postpartum, fever and infection, drug use such that would influence thermoregulation such as vasodilators, hemorrhage > 5 mL/kg, and patients who declined to participate.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were aged between 18-65 years and underwent surgery with general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Affect of two fresh gas flow rates (3lt/ 6lt min) on patients' airway temperature and humidity. | 2016-2018
  We will evaluate if different fresh gas flows effect on patients' airway temperature and moisture. We will evaluate by using a thermo-hygrometer fixed on anesthesia circuit.

SECONDARY OUTCOMES:
Affect of different anesthetic gases (sevoflurane, desflurane) and drugs (propofol)on patients' airway temperature and humidity. | 2016-2018
  We will evaluate if different anesthetic gases (sevoflurane, desflurane) and drugs (propofol) effect on patients' airway temperature and moisture. We will evaluate by using a thermo-hygrometer fixed on anesthesia circuit.

CONTACTS AND LOCATIONS:
Overall Officials: Ozkan Onal, Professor, Principal Investigator — Selcuk University

IPD SHARING:
Plan to Share IPD: Yes
The type(s) of supporting information that will be shared, in addition to the individual participant data set and data dictionaries for the IPD itself.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and any additional supporting information will become available in starting 2 months after publication.

REFERENCES:
- [Derived] Ozcan IG, Onal O, Ozdemirkan A, Saltali A, Sari M. Effects of different fresh gas flows and different anesthetics on airway temperature and humidity in surgical patients: a prospective observational study. Med Gas Res. 2022 Jul-Sep;12(3):83-90. doi: 10.4103/2045-9912.330691. PMID 34854418